CLINICAL TRIAL: NCT03388723
Title: The Role of Epigenetics in the Vicious Cycle of Diabetes and Pregnancy (VICYDIP)
Brief Title: Intergenerational Programming of Diabesity in Offspring of Women With Gestational Diabetes Mellitus
Acronym: InDiaGDM
Status: Completed | Type: Observational
Sponsor: Kem Hospital, Pune, India (Other)
Collaborators: Centre for Cellular and Molecular Biology, Hyderabad, India (Unknown)
Responsible Party: Principal Investigator, Dr. Chittaranjan S Yajnik, Director, Diabetes Unit, Kem Hospital, Pune, India
Other Study IDs: KEMHRC ID No. 1404
Record Dates: First submitted 2017-10-26; First posted 2018-01-03 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Gestational Diabetes
Keywords: Epigenetics; Cardiometabolic risk factors
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following biospecimens will be stored appropriately (at -80 degree C): Maternal blood in pregnancy, offspring's cord blood and placental tissue In the follow up study, samples from children born to diabetic and non diabetic mothers will be stored: blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1: Discovery phase: Approximately 150 women with Gestational Diabetes Mellitus (GDM) and 150 controls, and their offspring will be recruited in Pune (from KEM Hospital and Vadu). The objective will be:
  1. Identification of epigenetic signatures
  2. Measurements of B vitamins and 1-C metabolites in mothers' blood and cord blood
  3. Glucose, insulin and lipids in mothers during pregnancy
  4. Anthropometry and blood pressure
- Arm 2: Validation phase: Approximately 200 women with Gestational Diabetes Mellitus (GDM) and 200 controls, and their offspring will be recruited in Punjab, and 150 stored cord blood samples of GDM offspring in Pune will be investigated to validate the epigenetic signatures discovered in Arm 1.
- Arm 3: Stability phase: Approximately 500 offspring of women with Gestational Diabetes Mellitus (GDM) from Pune (~ half below 10 years and the rest over 10 years) will be investigated to study:
  1. Stability of epigenetic signatures in offspring through childhood and adolescence
  2. Relation of these signatures with phenotype

SUMMARY:
India is one of the diabetes capitals in the world. Indians are susceptible to develop diabetes at a younger age and at a lower BMI compared to Europeans. Current prevention strategies focus on reducing risk in those with the established disease or risk factors. The Developmental Origins of Health and Disease (DOHaD) hypothesis suggests that chronic non-communicable diseases (NCDs) are programmed by disturbances in maternal and fetal undernutrition. This offers an alternative primordial prevention strategy to reduce NCDs in future generations by improving health and nutrition of young women. Previous work in the Diabetes Unit, KEM Hospital, Pune has described the role of maternal micronutrients affecting 1-Carbon metabolism in the fetal programming of diabesity. In this application, the investigators offer to study other pathways of fetal programming i.e. maternal hyperglycemia and gestational diabetes mellitus (GDM) using an 'OMICs' approach. It is believed that epigenetic changes may be the main driver of programming. The investigators hypothesize that offspring of diabetic mothers will have different epigenetic signatures in cord blood and placenta compared to offspring of non-diabetic mothers. The investigators propose to study the effect of gestational hyperglycemia on newborn epigenetic signatures using the most appropriate technologies available and associate them with the underlying genotype. This will be performed on cord blood of 150 offspring of women with GDM and compared with a similar number of offspring of non-diabetic mothers recruited at Pune. The differentially methylated regions (DMRs) identified will then be validated by pyrosequencing in ~300 stored GDM cord blood samples in Pune. The investigators from Pune will also validate these markers in 200 newly recruited offspring of GDM and 200 controls from a different cohort in Punjab which has a different diet and lifestyle. The DMRs will also be validated in placental samples from both Pune and Punjab. The investigators will further test the stability of these markers and their associations with phenotype in a follow-up study of offspring of GDM mothers in upto 500 individuals. The investigators will compare the findings with the DNBC-GDM cohort in Denmark, allowing for differences in age, genetic make up, nutritional status and lifestyle. This study will help understand contribution of maternal diabetes to the current epidemic of diabesity and its molecular basis.

DETAILED DESCRIPTION:
The DOHaD paradigm proposes that early life nutrition and growth influence health and disease risk across the life-course. Intrauterine period is the most crucial period in these events, and contributes to fetal programming. Fetal undernutrition as well as over-nutrition (maternal obesity and diabetes) increase risk of diabetes in the offspring. Current thinking is that fetal programming is an 'epigenetic' phenomenon and the most prominent mechanism may be methylation of DNA and histones that regulate gene expression in key pathways. The investigators have previously highlighted a role for maternal micronutrients in fetal programming of adiposity, insulin resistance, and prediabetes (nutrient mediated teratogenesis). Now, the investigators propose to study the impact of maternal hyperglycemia during pregnancy on the future risk of diabesity in the offspring (fuel mediated teratogenesis). This programme, first of its kind in India, will undertake 'OMICs' measurements (DNA methylation and targeted metabolomics) on cord blood samples of children born to women with gestation diabetes mellitus (GDM), in studies in Pune, Western India (Arm-1) and Punjab, North India (Arm-2). Markers identified in the discovery phase will be investigated for validity and stability in blood, cord blood and placenta samples from children born to GDM mothers in the older cohorts in Pune and Punjab. Danish investigators will perform complimentary measurements in the Danish National Birth Cohort which will allow comparison of epigenetic markers in these two populations with widely different prevalence of GDM, and ethnic and nutritional factors. Special attention will be given to role of nutritional and lifestyle factors of mothers which influence the programming of fetal epigenome during pregnancy. The biobank of maternal, cord and offspring samples will be available in future to test newer hypotheses. This study will benefit from technology transfer across two countries. The findings will add substantially to the evidence base of intergenerational transmission of diabetes in a diabetic pregnancy, and will inform policy-makers to help curb the escalating epidemic of diabetes in India.

Hypotheses

1. The molecular mechanisms underlying the associations between gestational diabetes in the mother and diabesity in the offspring may involve permanent changes of DNA methylations in various tissues including blood cells obtained at birth and/or during childhood defining different trajectories.
2. Epigenetic fingerprints linking GDM with risk of T2D among the offspring may or may not be influenced by tissue of origin, diet, life-style and ethnicity of population.
3. Epigenetic changes in blood cells obtained at birth and/or during childhood associated with GDM in pregnancy may be used as bio-markers to predict later development of T2D in the offspring
4. The risk of developing diabetes among offspring of GDM women may be influenced by maternal factors operating during pregnancy including degree of hyperglycemia, obesity, dietary factors including composition of macro- and micronutrients, and/or by the level of physical activity of the mother.

ELIGIBILITY:
Inclusion Criteria:

Arm 1 and 2:

1. GDM or NGT on 75g OGTT (IADPSG Criteria).
2. Willing to participate and sign consent
3. Planned delivery at study site
4. Age > 18 years
5. Singleton pregnancy.

Arm 3:

1. Offspring of diabetic mothers and non diabetic mothers ( >2 years of age).

Exclusion Criteria:

Arm 1 and 2:

1. Severe medical/ surgical illness detrimental to pregnancy or delivery (Severe liver, renal, cardiovascular, pulmonary, hematologic, endocrine disorder or long term steroid use for any reason)
2. K/C/O Diabetes (Type 1 or Type 2 or any other type)
3. Severe anemia (Hemoglobin< 9 gm% in first trimester and < 8 gm% in second or third trimester)
4. IVF pregnancy.

Arm 3: None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Arm 1 and Arm 2: GDM women (diagnosed on OGTT) and women with normal glucose tolerance on OGTT and their offspring.
  Arm 3: Offspring of diabetic mothers and non diabetic mothers
Sampling Method: Non-Probability Sample
Enrollment: 1178 (Actual)
Dates: Start 2014-09-02 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Epigenetic signatures in the cord blood of the offspring of GDM mothers. | Upto 3 years from the start of the study
  The Illumina Infinium Human Methylation 450K array will be used for DNA methylation study. It generates a quantitative measurement of DNA methylation for >480,000 CpG sites spanning all annotated genes and other functional motifs. Markers influencing risk of diabetes and obesity will be of special interest. Approximately 150 GDM and 150 normal glucose tolerant pregnancies will contribute the samples.

SECONDARY OUTCOMES:
Association of the genotype with differentially methylated DNA regions. | Upto 3.5 years from the start of the study
  The Human OmniExpress Exome BeadChip will be used for generating genome wide data. It provides a backbone of >700,000 genome-wide markers (SNPs >5% minor allele frequencies) and 240,000 coding SNPs of all frequencies. This will allow to identify the variants that act as meQTLS.
Validation of the epigenetic signatures generated in Primary Outcome 1. | Upto 3.5 years from the start of the study
  Quantitative profile of DNA methylation at specific CpG sites will be done using Bisulfite Pyrosequencing [Sequenom EpiTYPER], in cord blood samples obtained in Pune and in Ludhiana.
Stability of epigenetic signatures discovered in the cord blood in offspring GDM mothers from childhood through adolescence. | Upto 4 years from the start of the study
  The cord blood differential epigenetic signatures will be investigated in the blood sample of the offspring of GDM mothers during childhood and adolescence. These children were born to GDM patients attending the diabetes clinic at KEM hospital, Pune over last 2 decades.
Association between epigenetic signatures and offspring phenotype at birth , and in childhood and adolescence. | Upto 4 years from the start of the study
  Following phenotype measures will be tested :
  1. Weight (Kg)
  2. Height (cm)
  3. BMI (Kg/m^2)
  4. Waist circumference (cm)
  5. Hip circumference (cm)
  6. Skinfolds (mm)
  7. DXA [ body composition measures: fat, lean and bone]
  8. Plasma Glucose concentration (mg/dl) in the cord blood and during an OGTT in childhood and adolescence.
  9. Plasma Insulin (mU/L) in the cord blood and during an OGTT in childhood and adolescence
  10. Glucose and insulin indices (HOMA measures) in 8, 9.
  11. Blood lipids (Cholesterol, HDL, LDL and Triglycerides) in the cord blood and during an OGTT in childhood and adolescence.
Qualitative and quantitative comparison of epigenetic signatures in the offspring of GDM mothers [Indian and Danish cohort]. | Upto 4.5 years from the start of the study
  Epigenetic signatures from Indian and Denmark cohorts will be compared, taking into account differences in genetic background, nutrition and lifestyle.
  Comparison will focus on the direction and strength of associations, and the metabolic pathways implicated in the above analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Chittaranjan Chittaranjan, MD FRCP, Principal Investigator — Director, Diabetes Unit, KEM Hospital Research Centre
Locations (1):
- KEM Hospital, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dabelea D, Pettitt DJ. Intrauterine diabetic environment confers risks for type 2 diabetes mellitus and obesity in the offspring, in addition to genetic susceptibility. J Pediatr Endocrinol Metab. 2001 Sep-Oct;14(8):1085-91. doi: 10.1515/jpem-2001-0803. PMID 11592564
- [Background] Petitt DJ, Bennett PH, Knowler WC, Baird HR, Aleck KA. Gestational diabetes mellitus and impaired glucose tolerance during pregnancy. Long-term effects on obesity and glucose tolerance in the offspring. Diabetes. 1985 Jun;34 Suppl 2:119-22. doi: 10.2337/diab.34.2.s119. PMID 3996763
- [Background] Gluckman PD, Hanson MA, Cooper C, Thornburg KL. Effect of in utero and early-life conditions on adult health and disease. N Engl J Med. 2008 Jul 3;359(1):61-73. doi: 10.1056/NEJMra0708473. No abstract available. PMID 18596274
- [Background] Wu L, Cui L, Tam WH, Ma RC, Wang CC. Genetic variants associated with gestational diabetes mellitus: a meta-analysis and subgroup analysis. Sci Rep. 2016 Jul 29;6:30539. doi: 10.1038/srep30539. PMID 27468700
- [Background] Ma RC, Tutino GE, Lillycrop KA, Hanson MA, Tam WH. Maternal diabetes, gestational diabetes and the role of epigenetics in their long term effects on offspring. Prog Biophys Mol Biol. 2015 Jul;118(1-2):55-68. doi: 10.1016/j.pbiomolbio.2015.02.010. Epub 2015 Mar 16. PMID 25792090
- [Background] Yajnik CS. Fetal programming of diabetes: still so much to learn! Diabetes Care. 2010 May;33(5):1146-8. doi: 10.2337/dc10-0407. No abstract available. PMID 20427687
- [Background] Kale SD, Yajnik CS, Kulkarni SR, Meenakumari K, Joglekar AA, Khorsand N, Ladkat RS, Ramdas LV, Lubree HG. High risk of diabetes and metabolic syndrome in Indian women with gestational diabetes mellitus. Diabet Med. 2004 Nov;21(11):1257-8. doi: 10.1111/j.1464-5491.2004.01337.x. No abstract available. PMID 15498096
- [Background] Kale SD, Kulkarni SR, Lubree HG, Meenakumari K, Deshpande VU, Rege SS, Deshpande J, Coyaji KJ, Yajnik CS. Characteristics of gestational diabetic mothers and their babies in an Indian diabetes clinic. J Assoc Physicians India. 2005 Oct;53:857-63. PMID 16459528
- [Background] Yajnik CS. Transmission of obesity-adiposity and related disorders from the mother to the baby. Ann Nutr Metab. 2014;64 Suppl 1:8-17. doi: 10.1159/000362608. Epub 2014 Jul 23. PMID 25059801